CLINICAL TRIAL: NCT04429126
Title: The Effect of Acupressure on Relieving Fatigue Following Traumatic Brain Injury: a Randomized Controlled Trial
Brief Title: Acupressure in Reducing Post-TBI Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associate Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109059-E
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4-point acupressure group (Experimental): The 5-point acupressure group will be instructed on the following acupressure points: sanyinjiao (SP6), Zu San Li (ST36), shenmen (TF4), Yongquan (KI-1), and He Gu (LI4).
  Bilateral 1.5 min for each point, three times daily for 4 weeks.
  Interventions: Behavioral: Acupressure
- 4 -point acupressure group (Active Comparator): The 2-point acupressure group will be instructed on the following acupressure points: He Gu (LI4) and Tai Chong (LV3).
  Bilateral 1.5 min for each point, three times daily for 4 weeks.
  Interventions: Behavioral: Acupressure
- Usual care (No Intervention): The usual care group will be required to maintain their daily activities. Weekly telephone follow-up will be conducted by principle investigator.

INTERVENTIONS:
Behavioral: Acupressure — Two types acupressure interventions, 5-point and 2-point acupressure groups, will be conducted in the current study.
  Arms: 4 -point acupressure group; 4-point acupressure group

SUMMARY:
Fatigue is a common symptom experienced by patients with traumatic brain injury (TBI). Prior works have demonstrated that it may profoundly impact the ability to return to productive activity and cognitive functions. However, few interventions have been applied in this population.The purpose of the current will be to test the effect of acupressure on fatigue reduction after traumatic brain injury.

DETAILED DESCRIPTION:
Fatigue is a pervasive and critical long-lasting symptom experienced by patients with traumatic brain injury (TBI) and can persist up to months or years after head injury. However, thus far, only few non-pharmacological interventions, such as mindfulness, are implemented in reducing fatigue in TBI survivors. Prior works have suggested that acupressure can significantly improve fatigue in different populations, such as cancers survivors and patients with hemodialysis. Therefore, we would like to test whether acupressure effectively improve fatigue after TBI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with traumatic brain injury over 6 months with initial GCS (admitted GCS) from 3-12.
* Aged between 20-65 years
* Are able to communicate in Chinese and Mandarin
* Are able to complete the questionnaires
* Complain of tiredness and cannot be restored even after a rest.
* No physical disability and visual impairment

Exclusion Criteria:

* With skin lesion
* had diagnosis of neuropathy and paraesthesia prior to study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigue | 4 weeks
  Self-reported feeling of tiredness, is measured by the Chinese version of The Mental fatigue Scale (MFS, higher scores indicate greater mental fatigue) and Multidimensional Fatigue Inventory (MFI, higher score indicates more fatigue)

SECONDARY OUTCOMES:
Memory function | 4 weeks
  The function will be measured by using the Rey Auditory Verbal Learning Test
Attention function | 4 weeks
  The function will be measured by using the Trail Making Test
Heart rate variability | My ECG E3-8010
  We will measure HRV parameter using the device of My ECG E3-8010
Brain waves | 4 weeks
  measured by the NeuroSky MindWave Mobile 2
Sleep quality | 4 weeks
  Sleep quality will be assessed by using the Pittsburgh Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yean Chiu, PhD, Principal Investigator — School of Nursing, Taipei Medical University
Locations (1):
- Hsiao-Yean Chiu, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No